CLINICAL TRIAL: NCT02694601
Title: Stimulate the Ketogenesis by Using a Caffeine Supplement
Brief Title: Ketone Production With Acute Caffeine Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-441
Record Dates: First submitted 2016-02-09; First posted 2016-02-29 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Healthy Adults
Keywords: Ketones; Glucose; Caffeine
MeSH Terms: conditions — Ketosis | interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketonemia following caffeine intake (Experimental): Participants have to follow three sequential visits of four hours each, which included a breakfast with one of the doses (2.5 or 5 mg/kg) of the caffeine supplement or without any supplement (baseline) and repeated blood sampling in order to evaluate ketone concentrations.
  Intervention 1: Control; no caffeine intake Intervention 2: Caffeine low dose (2.5 mg/kg of BW) Intervention 3: Caffeine high dose (5.0 mg/kg of MW)
  Interventions: Dietary Supplement: Control; Dietary Supplement: Caffeine low dose; Dietary Supplement: Caffeine high dose

INTERVENTIONS:
Dietary Supplement: Control — 4-hour visit with no caffeine is given during a standardize breakfast follow by repeated blood sampling.
  Other Names: CTL
Dietary Supplement: Caffeine low dose — 4-hour visit with a dose of 2.5 mg/kg of caffeine is given during a standardize breakfast follow by repeated blood sampling.
Dietary Supplement: Caffeine high dose — 4-hour visit with a dose of 5 mg/kg of caffeine is given during a standardize breakfast follow by repeated blood sampling.

SUMMARY:
Evaluate the effect of a caffeine supplement on the stimulation of lipolysis and the production of ketones in healthy adults (N=10).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of a caffeine supplement on the stimulation of lipolysis and the production of ketones in healthy adults (N=10). Two different doses of caffeine (2.5 mg/kg of BW and 5 mg/kg of BW) are compared. All the participants have to follow three sequential visits of four hours each, which included a breakfast with one of the doses (2.5 or 5 mg/kg) of the caffeine supplement or without any supplement (baseline) and repeated blood sampling in order to evaluate ketone concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* 18 years old and over

Exclusion Criteria:

* Drinking more than 300 mg of caffeine per day
* Diabetes or prediabetes
* Abnormal liver and kidney function
* Uncontrolled dyslipidemia, blood pressure
* Use of drugs known to influence the metabolism of lipids and carbohydrates (steroid, beta-blockers, diuretics, insulin sensitizer, etc.)
* Severe inflammation or infection
* Pregnancy
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, PhD, Principal Investigator — Research Centre on Aging - CSSS-IUGS - CIUSSS de l'Estrie - CHUS
Locations (1):
- Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketonemia Following Caffeine Intake: Participants have to follow three sequential visits of four hours each, which included a breakfast with one of the doses (2.5 or 5 mg/kg) of the caffeine supplement or without any supplement (baseline) and repeated blood sampling in order to evaluate ketone concentrations.
  Intervention 1: Control; no caffeine intake Intervention 2: Caffeine low dose (2.5 mg/kg of BW) Intervention 3: Caffeine high dose (5 mg/kg of BW)
Period: Overall Study
Arm/Group | Ketonemia Following Caffeine Intake
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketonemia Following Caffeine Intake
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Plasma Acetoacetate Concentrations
Description: Plasma acetoacetate (µmol/L) measured over a 4 hour period.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Ketonemia Following Caffeine Intake
Number analyzed (Participants) | 10
µmol/L
  CTL | 26.06 (3.71)
  Caffeine low dose | 30.99 (5.97)
  Caffeine high dose | 32.10 (8.40)

2. Primary Outcome: Plasma Beta-hydroxybutyrate Concentrations
Description: Plasma beta-hydroxybutyrate (µmol/L) measured over a 4 hour period.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Ketonemia Following Caffeine Intake
Number analyzed (Participants) | 10
µmol/L
  CTL | 92.69 (12.41)
  Caffeine low dose | 127.57 (16.98)
  Caffeine high dose | 144.99 (16.77)

3. Secondary Outcome: Plasma Glucose Concentrations
Description: Plasma glucose (mmol/L) measured over a 4 hour period.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Ketonemia Following Caffeine Intake
Number analyzed (Participants) | 10
mmol/L
  CTL | 4.95 (0.35)
  Caffeine low dose | 4.96 (0.29)
  Caffeine high dose | 4.98 (0.25)

4. Secondary Outcome: Plasma Cholesterol Concentrations
Description: Plasma cholesterol (mmol/L) measured over a 4 hour period.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Ketonemia Following Caffeine Intake
Number analyzed (Participants) | 10
mmol/L
  CTL | 4.26 (0.47)
  Caffeine low dose | 4.76 (0.35)
  Caffeine high dose | 4.81 (0.34)

5. Secondary Outcome: Plasma Triglyceride Concentrations
Description: Plasma triglycerides (mmol/L) measured over a 4 hour period.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Ketonemia Following Caffeine Intake
Number analyzed (Participants) | 10
mmol/L
  CTL | 0.90 (0.15)
  Caffeine low dosee | 0.92 (0.15)
  Caffeine high dosee | 0.97 (0.14)

ADVERSE EVENTS:
Time Frame: 3 visits of 4 hours
Groups:
- Ketonemia Following Caffeine Intake = Intervention 1: Control; no Caffeine Intake; Ketonemia Following Caffeine Intake = Intervention 2: Caffeine Low Dose (2.5 mg/kg of BW); Ketonemia Following Caffeine Intake = Intervention 3: Caffeine High Dose (5 mg/kg of BW): Participants have to follow three sequential visits of four hours each, which included a breakfast with one of the doses (2.5 or 5 mg/kg) of the caffeine supplement or without any supplement (baseline) and repeated blood sampling in order to evaluate ketone concentrations.
  Intervention 1: Control; no caffeine intake Intervention 2: Caffeine low dose (2.5 mg/kg of BW) Intervention 3: Caffeine high dose (5 mg/kg of BW)
Arm/Group | Ketonemia Following Caffeine Intake = Intervention 1: Control; no Caffeine Intake | Ketonemia Following Caffeine Intake = Intervention 2: Caffeine Low Dose (2.5 mg/kg of BW) | Ketonemia Following Caffeine Intake = Intervention 3: Caffeine High Dose (5 mg/kg of BW)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes